CLINICAL TRIAL: NCT00527046
Title: A Randomized, Double Blind, Placebo Controlled, Five Parallel Group Study Of The Effect Of CP-424,391 On Physical Performance And Body Composition In Older Subjects
Brief Title: Effects Of An Oral Growth Hormone Secretagogue In Older Functionally Limited Adults
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A257-102
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Aging; Frail Older Adults

INTERVENTIONS:
Drug: CP-424,391

SUMMARY:
A 24-month, placebo controlled, double dummy, parallel-design outpatient trial in generally healthy elderly men and women who are at risk of becoming frail.

ELIGIBILITY:
Inclusion Criteria:

65-84 years old, BMI < 30, at risk for functional decline based on SF-36, Instrumental Activities of Daily Living (per Nagy's), or 2 or more falls in prior 2 years

Exclusion Criteria:

Significant history or symptoms of acute medical conditions, currently in an exercise program, pain or other conditions that would prevent participating in exercise testing

Ages: 65 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 396 (Actual)
Dates: Start 1999-12; Primary Completion 2001-10 (Actual); Study Completion 2001-10 (Actual)

PRIMARY OUTCOMES:
Percent increase in lean (non fat) body mass. | Measured by DXA at BL 3, 6, 12, and 24 months
Change in functional performance (speed to climb stairs, walking speed and feet walked in 6 min). | Measured at BL, 3, 6, 12, and 24 months

SECONDARY OUTCOMES:
Pharmacokinetics, blood hormones and biomarkers | (BL,3,6,12,24 months)
Tape measurement of size of arm and leg muscles, waist, and hip | (BL,3,6,12,24 months)
IGF-1 and GH levels | (1,2,18 months)
Overnight GH profile in a subset | (2,18 months)
Muscle strength | (BL,3,6,12,24 months)
Questionnaires on general health, depression, mental status, sleep and activities of daily living | (BL,3,6,12,24 months)
Other physical performance tests including time to rise from a chair 5 times, balance tests (walking a straight line) | (BL,3,6,12,24 months)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (12):
- United States (12):
  - Pfizer Investigational Site, Palo Alto, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Hamden, Connecticut
  - Pfizer Investigational Site, New Britain, Connecticut
  - Pfizer Investigational Site, Lake Worth, Florida
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Seattle, Washington

REFERENCES:
- [Derived] White HK, Petrie CD, Landschulz W, MacLean D, Taylor A, Lyles K, Wei JY, Hoffman AR, Salvatori R, Ettinger MP, Morey MC, Blackman MR, Merriam GR; Capromorelin Study Group. Effects of an oral growth hormone secretagogue in older adults. J Clin Endocrinol Metab. 2009 Apr;94(4):1198-206. doi: 10.1210/jc.2008-0632. Epub 2009 Jan 27. PMID 19174493
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=102&StudyName=Effects+Of+An+Oral+Growth+Hormone+Secretagogue+In+Older+Functionally+Limited+Adults